CLINICAL TRIAL: NCT06469918
Title: The Co-Op @ HeartWorks
Status: Recruiting | Type: Observational
Sponsor: HeartWorks, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Co-Op 001
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Congenital Heart Disease
Keywords: HLHS; congenital heart defect; CHD; Hypoplastic left heart syndrome
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol is a research study involving human subjects diagnosed with Congenital Heart Defects/Disease (CHD). The Co-Op @ HeartWorks is a cooperative between the research platform at HeartWorks and members of the CHD community. Individuals choosing to participate will be referred to as 'members' of the co-op. This study aims to create a database of members medical journey data to inform future clinical innovation and design of clinical trials which address the needs of the members. The knowledge generated from this study will help advance the care of CHD patients through the deliberate action of The Co-Op @ HeartWorks members. Unlike a traditional disease registry, the members of The Co-Op @ HeartWorks will actively inform and contribute to the future studies affecting their health.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a congenital heart defects/disease
* Caregiver of a minor with a congenital heart defect/disease
* Authorized family member of a now deceased person with congenital heart defect/disease

Exclusion Criteria:

- Not having a congenital heart defect/disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Human subjects with congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2050-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Registry of individuals with CHD to plan and recruit for future interventional trials in Congenital Heart Defects/Disease | 25 years

CONTACTS AND LOCATIONS:
Locations (1):
- HeartWorks, Inc., Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

DOCUMENTS (1):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT06469918/Prot_000.pdf